CLINICAL TRIAL: NCT02852655
Title: A Pilot Surgical Trial To Evaluate Early Immunologic Pharmacodynamic Parameters For The PD-1 Checkpoint Inhibitor, Pembrolizumab (MK-3475), In Patients With Surgically Accessible Recurrent/Progressive Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Wen, MD, Patrick Wen, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-225
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Results first posted 2024-11-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Brain Cancer
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-surgery MK-3475 (Experimental): -After a screening phase of 14 days, eligible subjects will be randomized into two groups.
  * Pembrolizumab (MK3475) pre-surgery at pre-determine dosage followed by Pembrolizumab at pre-determine dosage every 3 weeks post surgery.
  * MK-3475 will be administered intravenously
  Interventions: Drug: MK-3475
- No MK-3475 at Pre-Surgery (Active Comparator): -After a screening phase of 14 days, eligible subjects will be randomized into two groups.
  * Pembrolizumab (MK-3475) at pre-determine dosage every 3 weeks post surgery.
  * MK-3475 will be administered intravenously
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475
  Other Names: Pembrolizumab

SUMMARY:
This research study is studying an immunotherapy as a possible treatment for Glioblastoma.

DETAILED DESCRIPTION:
PD-1 works to help tumor cells continue to grow and multiply. Pembrolizumab (MK-3475) is a humanized monoclonal antibody. Humanized monoclonal is an antibody that is designed to block the action of the receptor, PD-1.

The FDA (the U.S. Food and Drug Administration) has not approved Pembrolizumab for Glioblastoma but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma). Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made.
* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Have a Karnofsky performance status (KPS) ≥ 70 (Appendix A).
* Previous first line therapy with at least radiotherapy.
* Be at first or second relapse. Note: Relapse is defined as progression following initial therapy (i.e., radiation ± chemotherapy). For participants who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of registration.

Table 1 Adequate Organ Function Laboratory Values

* System Laboratory Value
* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
* Renal

  * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X institutional upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
  * Serum total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN OR ≤ 5 X institutional ULN for subjects with Gilberts syndrome
  * Albumin >2.5 mg/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT)
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

    ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Creatinine clearance should be calculated per institutional standard.
* CT or MRI within 14 days prior of registration.
* An interval of at least 4 weeks (to registration) between prior surgical resection or one week for stereotactic biopsy.
* An interval of at least 12 weeks from the completion of radiation therapy to registration unless there is unequivocal histologic confirmation of tumor progression.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* From registration, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies (including vaccines). No wash-out period required from TTF.
* Participants must have sufficient tissue from prior surgery revealing glioblastoma or variants for submission following registration. The following amount of tissue is required:

  * 1 formalin-fixed paraffin-embedded (FFPE) tumor tissue block (preferred) OR
  * 10 FFPE unstained slides (5 μm thick)
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers. Patients must be eligible for surgical resection with the expectation that the surgeon is able to resect at least 400mg of tumor with low risk of inducing neurological injury.
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must agree to use highly effective contraception during study treatment and for 120 days after study discontinuation. Highly effective contraception is defined as either:

  * True Abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Sterilization: Surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment (as described in item 3.1.16 above).
  * Male Partner Sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner must be the sole partner for that participant.
  * Use of a combination of any two of the following:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    * Appropriate hormonal contraceptives (including any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent - including oral, subcutaneous, intrauterine, or intramuscular agents)
* Male subjects must agree to use adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy.

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency.
* Has tumor primarily localized to the brainstem or spinal cord.
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc) within six months of registration.
* Has received anti-angiogenic or anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc).
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 4 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of registration.
* Has received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or convection enhanced delivery.
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of registration.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of registration.
* Has a known additional malignancy that is progressing or requires active treatment within 3 years of registration. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Examples include but are not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to registration.
* Has a known hypersensitivity to any of the study therapy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer, New York, New York
  - UT, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFaline-Figueroa JR, Sun L, Youssef GC, Huang R, Li G, Kim J, Lee EQ, Nayak L, Chukwueke U, Beroukhim R, Batchelor TT, Chiocca EA, Everson RG, Doherty L, Stefanik J, Partridge K, Spearman A, Myers A, Westergaard C, Russ A, Lavallee M, Smokovich A, LaForest-Roys C, Garcia Fox R, McCluskey C, Bi WL, Arnaout O, Peruzzi P, Cosgrove GR, Ligon KL, Arrillaga-Romany I, Clarke JL, Reardon DA, Cloughesy TF, Prins RM, Wen PY. Neoadjuvant anti-PD1 immunotherapy for surgically accessible recurrent glioblastoma: clinical and molecular outcomes of a stage 2 single-arm expansion cohort. Nat Commun. 2024 Dec 30;15(1):10757. doi: 10.1038/s41467-024-54326-7. PMID 39737895

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Stage 1): Neoadjuvant + Adjuvant MK3475; Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475: * Single dose of Pembrolizumab (MK3475) @ 200 mg IV
  * Surgery within 14 days (+/- 5 days) of Neoadjuvant dose
  * Adjuvant Pembrolizumab (MK3475) @ 200 mg IV every 3 weeks to start upon recovery from surgery (and no more than 35 days after surgery) until disease progression or unacceptable toxicity.
  * Pembrolizumab (MK-3475) administered intravenously over 30 minutes (-5 min/+10 min)
- Group B (Stage 1): Adjuvant MK3475: * Surgery (NO pre-surgical drug)
  * Adjuvant Pembrolizumab (MK3475) @ 200 mg IV every 3 weeks to start upon recovery from surgery (and no more than 35 days after surgery) until disease progression or unacceptable toxicity.
  * Pembrolizumab (MK-3475) administered intravenously over 30 minutes (-5 min/+10 min)
Period: Registered and Ready to Initiate Tx
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475
Started | 16 | 25 | 19
Completed | 16 | 25 | 16
Not Completed | 0 | 0 | 3
Not completed — Patient deemed ineligible due to high decadron dose | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Period: Receive NeoAdjuvant Protocol Tx
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475
Started | 16 | 25 | 16
Completed | 16 | 25 | 16
Not Completed | 0 | 0 | 0
Period: Complete Surgical Resection
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475
Started | 16 | 25 | 16
Completed | 16 | 25 | 16
Not Completed | 0 | 0 | 0
Period: Eligible to Initiate Adjuvant MK3475
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475
Started | 16 | 25 | 16
Completed | 15 | 22 | 14
Not Completed | 1 | 3 | 2
Not completed — Disease Progression | 1 | 2 | 2
Not completed — Surgery showed no evidence of recurrence (only treatment related changes) | 0 | 1 | 0
Period: Adjuvant MK3475 Therapy
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475
Started | 15 | 22 | 14
Completed | 0 | 0 | 0
Not Completed | 15 | 22 | 14
Not completed — Disease Progression | 13 | 21 | 12
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Still on Active Study Therapy | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Stage 1): Neoadjuvant + Adjuvant MK3475 | Group A Expansion Cohort (Stage 2): Neoadjuvant + Adjuvant MK3475 | Group B (Stage 1): Adjuvant MK3475 | Total
Number analyzed (Participants) | 16 | 25 | 16 | 57
Age, Customized [Number; unit: years]
  21-29 years old | 1 | 1 | 0 | 2
  30-39 years old | 2 | 2 | 2 | 6
  40-49 years old | 1 | 6 | 0 | 7
  50-59 years old | 3 | 3 | 5 | 11
  60-69 years old | 9 | 10 | 6 | 25
  70 + | 0 | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 11 | 26
  Male | 9 | 17 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 13 | 21 | 13 | 47
  Unknown or Not Reported | 1 | 3 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 15 | 18 | 12 | 45
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 6 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 16 | 25 | 16 | 57
Baseline Karnofsky Performance Status (KPS) [Number; unit: participants] — KPS performance scale (0-100):
  * 100 - Normal, no complaints; no evidence of disease.
  * 90 - Able to carry on normal activity; minor signs or symptoms of disease.
  * 80 - Normal activity with effort; some signs or symptoms of disease.
  * 70 - Cares for self; unable to carry on normal activity or to do active work.
  participants
    KPS = 70 | 5 | 2 | 1 | 8
    KPS = 80 | 7 | 9 | 4 | 20
    KPS = 90 | 3 | 14 | 11 | 28
    KPS = 100 | 1 | 0 | 0 | 1
Current Relapse # [Count of Participants; unit: Participants]
  1st Relapse | 12 | 24 | 15 | 51
  2nd Relapse | 4 | 1 | 1 | 6
Total Daily Steroid Dose at Registration (mg/day) [Count of Participants; unit: Participants]
  0 mg/day | 9 | 20 | 9 | 38
  1 mg/day | 2 | 0 | 1 | 3
  2 mg/day | 2 | 1 | 2 | 5
  3 mg/day | 1 | 0 | 0 | 1
  4 mg/day | 2 | 4 | 3 | 9
  6 mg/day | 0 | 0 | 1 | 1
MGMT Methylation Status [Count of Participants; unit: Participants]
  MGMT Methylated | 6 | 12 | 11 | 29
  MGMT Unmethylated | 7 | 11 | 4 | 22
  Unknown | 3 | 2 | 1 | 6
IDH1/2 Mutation Status [Count of Participants; unit: Participants]
  Negative | 12 | 24 | 13 | 49
  Positive | 3 | 1 | 2 | 6
  Unknown | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Infiltrating T Lymphocyte (TIL) Density
Description: To measure changes in tumor infiltrating T lymphocyte (TIL) density, defined as % total cells. It will be assessed using pooled Group A and Group B patients.
Time Frame: 2 weeks. TIL density is determined in surgical tumor tissue; on-study surgery occurs 14 days (+/- 5 days) after Neoadjuvant Day 1.
Population: Group A = Initial Group A Cohort (Stage 1) + Group A Expansion Cohort (Stage 2) Group B = Initial Group B Cohort (Stage 1)
Measure: Mean (Standard Error); unit: percentage of total stromal area
Groups:
- Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort): * Single dose of Pembrolizumab (MK3475) @ 200 mg IV
  * Surgery within 14 days (+/- 5 days) of Neoadjuvant dose
  * Adjuvant Pembrolizumab (MK3475) @ 200 mg IV every 3 weeks to start upon recovery from surgery (and no more than 35 days after surgery) until disease progression or unacceptable toxicity.
  * Pembrolizumab (MK-3475) administered intravenously over 30 minutes (-5 min/+10 min)
- Group B: Adjuvant MK3475 (Stage 1 Cohort): * Surgery (NO pre-surgical drug)
  * Adjuvant Pembrolizumab (MK3475) @ 200 mg IV every 3 weeks to start upon recovery from surgery (and no more than 35 days after surgery) until disease progression or unacceptable toxicity.
  * * Pembrolizumab (MK-3475) administered intravenously over 30 minutes (-5 min/+10 min)
Arm/Group | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) | Group B: Adjuvant MK3475 (Stage 1 Cohort)
Number analyzed (Participants) | 37 | 15
percentage of total stromal area | 2.2 (0.32) | 2.1 (0.63)

2. Primary Outcome: Cell Cycle and Cancer Proliferation Genetic Signature
Description: To measure changes in cell cycle and cancer proliferation genetic signature; these results are reported using Gene Set Variation Analysis (GSVA) absolute enrichment scores (ES). GSVA scores are unit-less scores derived by comparing mRNA expression of a specific gene set to genes outside of the gene set in a sample. In this case, GSVA scores for "Farmers_breast_cancer_cluster_2, as previously described" were utilized.
  PMID 30742122 (https://pubmed.ncbi.nlm.nih.gov/30742122/) and PMID 23323831 (https://pubmed.ncbi.nlm.nih.gov/23323831/)
  It will be assessed using pooled Group A and Group B patients.
Time Frame: 2 weeks. Cell cycle/cancer proliferation genetic signature is determined in surgical tumor tissue; on-study surgery occurs 14 days (+/- 5 days) after Neoadjuvant Day 1.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) | Group B: Adjuvant MK3475 (Stage 1 Cohort)
Number analyzed (Participants) | 34 | 15
unitless | -0.1758 (0.08192) | 0.3008 (0.1472)

3. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Number of Participants who Experienced a Serious Adverse Event (SAE) or Event of Clinical Interest (ECI) Deemed At Least Possibly Related to Pembrolizumab (MK3475). The following are measured as part of safety: laboratory safety assessments, KPS status, vital signs and physical examinations.
Time Frame: 5 years. Although there is still 1 patient on active study treatment as of today (4/1/2024), we stopped looking at this information as of 6/2/2022 for study reporting purposes.
Population: All patients who received at least one dose of pembrolizumab on study are included in this analysis.
  Group A = Initial Group A Cohort (Stage 1) + Group A Expansion Cohort (Stage 2) Group B = Initial Group B Cohort (Stage 1)
Measure: Count of Participants; unit: Participants
Groups:
- Group B: Adjuvant MK3475 (Stage 1 Cohort): * Surgery (NO pre-surgical drug)
  * Adjuvant Pembrolizumab (MK3475) @ 200 mg IV every 3 weeks to start upon recovery from surgery (and no more than 35 days after surgery) until disease progression or unacceptable toxicity.
  * Pembrolizumab (MK-3475) administered intravenously over 30 minutes (-5 min/+10 min)
Arm/Group | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) | Group B: Adjuvant MK3475 (Stage 1 Cohort)
Number analyzed (Participants) | 41 | 16
Participants
  Patients Experiencing an SAE Deemed At Least Possibly Related to Pembrolizumab | 13 | 5
  Patients Experiencing an ECI Deemed At Least Possibly Related to Pembrolizumab | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: To determine the efficacy of pembrolizumab in patients with surgically accessible recurrent/progressive glioblastoma (GBM) participants as measured by 6-month progression-free survival (PFS6) using Radiologic Assessment in Neuro-Oncology (RANO) criteria.
  Progression is defined using RANO criteria, as any of the following:
  1. ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement, on stable or increasing doses of corticosteroids
  2. Any new enhancing measurable lesion
  3. Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose
  4. Or failure to return for evaluation as a result of death or deteriorating condition
Time Frame: 180 Days
Population: Censoring & Final PFS #s:
  • Group A patients censored from PFS Analysis:
  o 1 patient's on study surgery did not show recurrent disease (53)
  Group A = Initial Stage 1 Cohort + Stage 2 Expansion Cohort Group B = Initial Stage 1 Cohort
  * 1 patient's histology did not confirm diagnosis of GBM (28)
  * 3 patients' disease was considered unevaluable (47, 49, & 60)
    • Group B patients censored from PFS Analysis:
  * 1 patient's on study surgery did not show recurrent disease (13)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) | Group B: Adjuvant MK3475 (Stage 1 Cohort)
Number analyzed (Participants) | 36 | 15
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) on this trial have been monitored/assessed for up to 6 years (the maximum amount of time a patient has remained on active study treatment). AEs are collected from the time of treatment registration through 30 days following end of study treatment. AEs meeting serious criteria, from the time of consent through 90 days following end of study treatment, or initiation of new anti-cancer therapy, whichever is earlier.
Description: An AE is any untoward medical occurrence in a subject receiving study treatment, regardless of event causality. An SAE is an AE at any dose that: results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, is a new cancer, is associated with an overdose, or is an important medical event. One Group A subject was lost-to-follow-up, so was tracked for a shorter duration.
Arm/Group | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) | Group B: Adjuvant MK3475 (Stage 1 Cohort)
All-Cause Mortality (participants affected / at risk) | 37/41 | 16/16
Serious Adverse Events (participants affected / at risk) | 18/41 | 9/16
Other Adverse Events (participants affected / at risk) | 40/41 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) (N=41) | Group B: Adjuvant MK3475 (Stage 1 Cohort) (N=16)
Sinus tachycardia (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 1
Gait disturbance (General disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 5 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 5 | 1
Confusion (Psychiatric disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify: Failure to Thrive (General disorders) | 1 | 0
Vulval infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lethargy (Nervous system disorders) | 2 | 0
Nervous system disorders - Other, specify: Left-sided neglect (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Surgical and medical procedures - Other, specify: Craniotomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Neoadjuvant + Adjuvant MK3475 (Stage 1 Cohort + Stage 2 Expansion Cohort) (N=41) | Group B: Adjuvant MK3475 (Stage 1 Cohort) (N=16)
Anemia (Blood and lymphatic system disorders) | 16 | 7
Sinus bradycardia (Cardiac disorders) | 5 | 1
Sinus tachycardia (Cardiac disorders) | 7 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 7 | 1
Hypothyroidism (Endocrine disorders) | 10 | 0
Blurred vision (Eye disorders) | 2 | 1
Dry eye (Eye disorders) | 1 | 1
Optic nerve disorder (Eye disorders) | 5 | 1
Scleral disorder (Eye disorders) | 0 | 1
Eye disorders - Other, specify: Double Vision (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 6 | 6
Diarrhea (Gastrointestinal disorders) | 10 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 8
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 3
Edema face (General disorders) | 3 | 2
Edema limbs (General disorders) | 4 | 0
Edema trunk (General disorders) | 0 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 18 | 12
Fever (General disorders) | 0 | 3
Gait disturbance (General disorders) | 15 | 4
Localized edema (General disorders) | 4 | 1
Malaise (General disorders) | 3 | 2
Pain (General disorders) | 4 | 1
Sinusitis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Propionibacterium acnes - CNS (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 8 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 10 | 2
Alkaline phosphatase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 2
Blood bilirubin increased (Investigations) | 1 | 2
Cholesterol high (Investigations) | 3 | 0
Creatinine increased (Investigations) | 6 | 0
INR increased (Investigations) | 4 | 1
Lymphocyte count decreased (Investigations) | 14 | 9
Lymphocyte count increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 4
Platelet count decreased (Investigations) | 9 | 5
Weight gain (Investigations) | 3 | 0
White blood cell decreased (Investigations) | 8 | 5
Anorexia (Metabolism and nutrition disorders) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 5
Hypokalemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 10 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 11 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Ataxia (Nervous system disorders) | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 2
Cognitive disturbance (Nervous system disorders) | 7 | 2
Concentration impairment (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 10 | 4
Dysarthria (Nervous system disorders) | 5 | 2
Dysesthesia (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Dysphasia (Nervous system disorders) | 5 | 4
Edema cerebral (Nervous system disorders) | 9 | 1
Facial muscle weakness (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 23 | 9
Intracranial hemorrhage (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 10 | 3
Movements involuntary (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 6 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2
Seizure (Nervous system disorders) | 13 | 3
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 3 | 2
Nervous system disorders - Other, specify: Tumor Flair (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify: left slowed finger tapping (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify: Left pronator drift (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify: left visual field cut (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 7 | 2
Confusion (Psychiatric disorders) | 10 | 1
Depression (Psychiatric disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 4 | 5
Personality change (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 5 | 1
Urinary urgency (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory, thoracic and mediastinal disorders, Other: Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 3 | 0
Surgical and medical procedures - Other, specify: IVC filter placement (Surgical and medical procedures) | 1 | 1
Hypertension (Vascular disorders) | 10 | 1
Hypotension (Vascular disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT02852655/Prot_SAP_000.pdf